CLINICAL TRIAL: NCT03349866
Title: A Prospective Study of Apatinib Plus Concurrent Neoadjuvant Chemoradiotherapy for Siewert II ，III of Locally Advanced HER-2 Negative Adenocarcinoma at Gastroesophageal Junction
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hebei Medical University (Other)
Responsible Party: Principal Investigator, Qun Zhao, Principal Investigator, Hebei Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HRA-G01
Record Dates: First submitted 2017-11-17; First posted 2017-11-22 (Actual); Last update posted 2020-02-19 (Actual); Status verified 2020-02

CONDITIONS: Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — apatinib; Capecitabine; Oxaliplatin; Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- apatinib XELOX and radiotherapy (Experimental): apatinib：250mg qd po XELOX：Capecitabine 1000mg/m2 bid d1-14，Oxaliplatin 130 mg/m2 Ivgtt d1 q3w Radiotherapy：45Gy/25f （1.8Gy/f/d，5 f/w）
  Interventions: Drug: apatinib; Drug: Capecitabine; Drug: Oxaliplatin; Radiation: Radiotherapy
- XELOX and radiotherapy (Active Comparator): XELOX：Capecitabine 1000mg/m2 bid d1-14，Oxaliplatin 130 mg/m2 Ivgtt d1 q3w Radiotherapy：45Gy/25f （1.8Gy/f/d，5 f/w）
  Interventions: Drug: Capecitabine; Drug: Oxaliplatin; Radiation: Radiotherapy

INTERVENTIONS:
Drug: apatinib — apatinib：250mg qd po
  Arms: apatinib XELOX and radiotherapy
Drug: Capecitabine — 1000mg/m2 bid d1-14
Drug: Oxaliplatin — 130 mg/m2 Ivgtt d1 q3w
Radiation: Radiotherapy — 45Gy/25f （1.8Gy/f/d，5 f/w）

SUMMARY:
The purpose of this study is to assess the efficacy and safety of patients who receive concurrent neoadjuvant chemoradiotherapy for Siewert II ，III of locally advanced HER-2 negative adenocarcinoma at gastroesophageal junction.

ELIGIBILITY:
Inclusion Criteria:

1. Age:18 to 70 years old (man or female);
2. Conﬁrmed to Siewert II , III of locally advanced adenocarcinoma at gastroesophageal junction and tumor long diameter ≤8 cm by gastroscopy and CT, The her-2 negative was detected by immunohistochemistry;
3. Patients with Stage for Ⅲ by CT/MRI (According to the eighth edition of AJCC );
4. Patients with measurable lesions(measuring≥10mm on spiral CT scan, satisfying the criteria in RECIST1.1);
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1;
6. Major organ function has to meet the following certeria:

   HB≥80g/L; ANC≥1.5×109/L; PLT≥90×109/L; ALT and AST≤2.5×ULN, but<≤5×ULN if the transferanse elevation is due to liver metastases； TBIL<1.5×ULN； Serum creatinine ≤1.5×ULN;
7. Life expectancy greater than or equal to 6 months;
8. Women of childbearing age must have contraceptive measures or have test pregnancy (serum or urine) enroll the study before 7 days, and the results must be negative, and take the methods of contraception during the test and the last to have drugs after 8 weeks. Men must be contraception or has sterilization surgery during the test and the last to have drugs after 8 weeks;
9. Participants were willing to join in this study, and written informed consent, good adherence, cooperate with the follow-up.

Exclusion Criteria:

1. Allergic to apatinib, capecitabine and oxaliplatin;
2. The cytological examination of the abdominal cavity washing fluid showed that the tumor shedding cells were positive;
3. Have high blood pressure and antihypertensive drug treatment can not control (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg), Uncontrolled coronary heart disease and arrhythmia ,classⅢ-Ⅳcardiac insufficiency;
4. A variety of factors influencing oral drugs (such as unable to swallow, nausea, vomiting, chronic diarrhea and intestinal obstruction, etc);
5. Patients with tendency of gastrointestinal bleeding, including the following: a local active ulcerative lesions, and defecate occult blood (+ +); Has melena and hematemesis in two months;
6. Coagulant function abnormality (INR > 1.5 ULN, APTT > 1.5 ULN), with bleeding tendency;
7. Pregnant or lactating women;
8. Patients with other malignant tumors within 5 years (except for curable skin basal cell carcinoma and cervical carcinoma in situ);
9. History of psychiatric drugs abuse and can't quit or patients with mental disorders;
10. Less than 4 weeks from the last clinical trial;
11. The researchers think inappropriate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2017-11-30 (Actual); Primary Completion 2019-11-30 (Actual); Study Completion 2020-11-30 (Estimated)

PRIMARY OUTCOMES:
The pathological complete response rate(pCR) | within 3 weeks after surgery
  The lesion disappeared completely by pathology

SECONDARY OUTCOMES:
Objective response rate (ORR) | within 3 weeks after surgery
  Baseline to measured stable disease
R0-resection rate | within 3 weeks after surgery
  There was no residual by the microscope
Disease-free survival(DFS) | 3 year
  Baseline to measured date of recurrence or death from any cause
Overall survival (OS) | 3years
  Baseline to measured date of death from any cause
Adverse events | 3 year
  Toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.The number of Participants with adverse events will be recorded at each treatment visit.

CONTACTS AND LOCATIONS:
Overall Officials: Qun Zhao, Principal Investigator — Hebei Medical University Fourth Hospital; Jun Wang, Principal Investigator — Hebei Medical University Fourth Hospital
Locations (1):
- The Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China

REFERENCES:
- [Derived] Guo H, Li Y, Lin C, Cheng Y, Zhang Z, Wang D, Zhao X, Liu Y, Jing S, Yang P, Tian Y, Liu Y, Wang J, Zhao Q. Efficacy and safety of neoadjuvant chemoradiotherapy plus apatinib for patients with locally advanced, HER2-negative, Siewert's type II-III adenocarcinoma of esophagogastric junction: a single-arm, open-label, phase II trial. Am J Transl Res. 2021 Aug 15;13(8):9015-9023. eCollection 2021. PMID 34540013